CLINICAL TRIAL: NCT02200185
Title: Efficacy and Safety of Nebulized Morphine Given at Two Different Doses Compared to Intravenous Morphine in Post-traumatic Acute Pain: a Randomized Controlled Double Blind Study
Brief Title: Titrated Versus High and Low Dose Nebulized Morphine to Reduce Pain in Emergency Settings
Acronym: TIMORNEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIMORNEB
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Post-Traumatic Headache; Acute Pain
Keywords: post traumatic pain; titrated morphine; nebulised morphine
MeSH Terms: conditions — Post-Traumatic Headache; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IV titrated morphine (Placebo Comparator): patient will receive 2 mg morphine each 5 min, associated to continuous nebulisation of saline serum (placebo).
  Morphine administration is stopped when VAS becomes under 50% and treatment failure is defined as VAS > 50%, 30 minutes after the beginning of the protocol.
  Interventions: Drug: IV titrated morphine
- Low dose nebulised morphine (Experimental): patient will receive 10 mg of morphine prepared with 4 ml saline serum (SS) and nebulised with 6 l/min flow during 10 minutes.
  Nebulisation will be repeated 3 times, in addition, patients receive 2 ml IV SS every 5 minutes as placebo
  Interventions: Drug: Low dose nebulised morphine
- High dose nebulised morphine (Experimental): patient will receive 20 mg of morphine prepared with 3 ml saline serum (SS) and nebulised with 6 l/min flow during 10 minutes.
  Nebulisation will be repeated 3 times, in addition, patients receive 2 ml IV SS every 5 minutes as placebo.
  Interventions: Drug: High dose nebulised morphine

INTERVENTIONS:
Drug: IV titrated morphine — Intravenous morphine : 2 mg every 5 minutes by IV root and nebulized placebo:
  * SS nebulised : 5 ml SS nebulised over 10 minutes and repeated 3 times
  Other Names: IV morphine group
  Arms: IV titrated morphine
Drug: Low dose nebulised morphine — 10 mg morphine in 4 ml Serum Saline(SS) nebulised over 10 minutes and repeated 3 times, and SS IV placebo : 2 ml by IV root every 5 minutes
  Other Names: Neb10
  Arms: Low dose nebulised morphine
Drug: High dose nebulised morphine — 20 mg morphine in 3 ml serum saline (SS) nebulised over 10 minutes and repeated 3 times, and SS IV placebo : 2 ml by IV root every 5 minutes
  Other Names: Neb20
  Arms: High dose nebulised morphine

SUMMARY:
The investigators test a different technique using morphine to improve pain relief in patient visiting the emergency department with acute trauma pain, for this we are comparing three different methods of morphine administration:

* intravenous titrated morphine
* low dose nebulized morphine and
* high dose nebulized morphine

DETAILED DESCRIPTION:
Trauma patients are frequent in emergency department settings, and often require urgent care.

taking care of this patients consists on taking care of their pain and then the specific treatment of their traumatic lesions.

actually, the most used medicine and most efficient one in treating pain is morphine, it's mechanism of action is by acting on receptors located on neuronal cell membranes and inhibit neurotransmitter release.

The most applied administration root of morphine is by intravenous (IV) titration or IV continuous perfusion, but until now, there is no clear recommendation concerning the superiority of this root over other administration techniques such as nebulization.

In this study we aimed to investigate the efficiency, the feasibility and the tolerance of three morphine administration roots in patients with acute traumatic pain and to clarify the most adequate one to apply in emergency department settings.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 8 years and less than 50 years
* patients who consult emergency department for sever pain after an immediately trauma

Exclusion Criteria:

* Glasgow coma scale <14
* inability to cooperate
* hypotension with systolic blood pressure< 90mmhg
* bradypnea<12cpm
* SAO2<90%
* polytrauma
* nasal trauma
* rhinitis
* nasal obstruction
* allergy to opioids

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain resolution | 30 minutes
  primary end point defined by the decrease in intensity pain objectified by a decline in visual analogy pain scale greater than or equal to 50% of its initial value

SECONDARY OUTCOMES:
side effects | 30 minutes
  secondary outcomes combine the occurrence of side effects requiring discontinuation of treatment such as: dizziness, dyspnea, cutaneous rush, vomiting, nausea and pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency Department, Monastir, Monastir Governorate, Tunisia

REFERENCES:
- [Derived] Grissa MH, Boubaker H, Zorgati A, Beltaief K, Zhani W, Msolli MA, Bzeouich N, Bouida W, Boukef R, Nouira S. Efficacy and safety of nebulized morphine given at 2 different doses compared to IV titrated morphine in trauma pain. Am J Emerg Med. 2015 Nov;33(11):1557-61. doi: 10.1016/j.ajem.2015.06.014. Epub 2015 Jun 14. PMID 26143313
- See also: official department site — http://www.urgencemonastir.com